CLINICAL TRIAL: NCT01970020
Title: An Open-Label Study to Investigate the Absorption, Metabolism, and Excretion of JNJ-38518168 in Healthy Subjects Following a Single Oral Dose Administration of 14C-JNJ-38518168
Brief Title: A Study to Investigate the Absorption, Metabolism, and Excretion of JNJ-38518168 After a Single Oral Dose in Healthy Male Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100989; 38518168ARA1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: Healthy; JNJ-38518168; 14C-JNJ-38518168; Absorption; Metabolism; Excretion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JNJ-38518168 (Experimental)
  Interventions: Drug: JNJ-38518168

INTERVENTIONS:
Drug: JNJ-38518168 — Following an at least 10-hour overnight fast, participants will receive a single dose containing 30 mg of 14C JNJ-38518168 given as an oral solution on Day 1

SUMMARY:
The purpose of the study is to investigate the absorption, metabolism, and excretion of 14C JNJ-38518168 in healthy adult male participants after a single oral dose of 30 mg 14C JNJ-38518168.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-center, single-arm (single group), and single-dose study. This study will include a screening period of 21 days prior to study medication administration. Six men will be enrolled and admitted to the clinical study unit on the morning of Day -1. On Day 1, participants will receive a single oral solution dose containing 30 mg of 14C JNJ-38518168 given as an oral solution. The participants will be confined to the clinical study unit for at least 360 hours after dosing ie, Day -1 through Day 14 and they will be discharged on Day 15; however, participants who, by Day 15, do not meet the discharge criteria will extend their residency in the study unit for up to Day 21. They will return to the study center 7 to 10 days after discharge for the final safety follow-up. The study will include the following safety evaluations: adverse event, vital sign, 12-lead electrocardiography, physical examination, and clinical laboratory test. For each participant the total duration in the study is approximately 6 weeks (including screening and safety follow-up) or 7 weeks for participants who extend the residence up to Day 21.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male participants with a body mass index 18 to 30 kg/m2 (inclusive) and a body weight not less than 50 kg
* Must use adequate contraception and not donate sperm during study and for 90 days after receiving the study medication
* Non-smoker and blood pressure between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic
* Have a 12-lead ECG consistent with normal cardiac conduction and function at screening

Exclusion Criteria:

* Exposure to radiation for professional or medical reasons in the past 12 months
* Recent changes in bowel habits (frequency, consistency, and amount) and irregular defecation pattern (less than one defecation per day)
* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease and coagulation disorders
* History of malignancy within 5 years before screening
* Has received a Bacille Calmette-Guérin vaccination within 12 months or any other live bacterial or live viral vaccination within 12 weeks prior to the first administration of study agent

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration of 14C JNJ-38518168 in plasma | Predose; and at 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, and 336 hours post-dose
Time to reach the maximum observed concentration of 14C JNJ-38518168 in plasma | Predose; and at 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, and 336 hours post-dose
Area under the concentration-time curve | Predose; and at 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, and 336 hours post-dose
Amount of 14C JNJ-38518168 excreted into the urine during a collection interval | Predose and from 0- to 4, 4- to 8, 8- to 12, 12- to 24, 24- to 36, 36- to 48 hours after dosing, and every 24 hours (pooled for 24-hour interval) thereafter until 336 hours post-dose
  Amount excreted into the urine during a collection interval, where t1 and t2 are the start and end times of the collection interval, and calculated by multiplying the urinary volume with the urinary concentration for that interval.
Amount of 14C JNJ-38518168 excreted into the feces during a collection interval | From Day -1 through Day 14
  Amount excreted into the feces during a collection interval, where t1 and t2 are the start and end times of the collection interval, and calculated by multiplying the feces weight with the feces concentration for that interval
Amount excreted into the vomit during a collection interval (applicable only for participants who experience vomitting) | Within 24 hours after dosing
  Amount excreted into the vomit during a collection interval, where t1 and t2 are the start and end times of the collection interval, and calculated by multiplying the weight of the vomit with the vomit concentration for that interval

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium